CLINICAL TRIAL: NCT03344874
Title: Comparison of Stethee® to the Conventional Stethoscope for Auscultation of Simulated Heart Sounds: A Randomised, Crossover, Non-Inferiority Trial (STELIT)
Brief Title: Comparison of Stethee® to the Conventional Stethoscope for Auscultation of Simulated Heart Sounds
Acronym: STELIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: M3DICINE Inc. (Other)
Responsible Party: Principal Investigator, Amanda Wei Yin Lim, Research Pharmacist, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: STELIT
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Heart Diseases
Keywords: heart sounds; Stethee; electronic stethoscope
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stethee (new stethoscope) (Experimental): Test 1: Use Stethee® to auscultate and identify a set of 10 manikin-simulated heart sounds.
  Test 2: After a 10-minute break, use 3MTM Littmann® Classic IIITM to auscultate and identify the same set of 10 manikin-simulated heart sounds but played in a different sequence to Test 1.
  Interventions: Device: Stethee®; Device: 3MTM Littmann® Classic IIITM
- Littmann (conventional stethoscope) (Active Comparator): Test 1: Use 3MTM Littmann® Classic IIITM to auscultate and identify a set of 10 manikin-simulated heart sounds.
  Test 2: After a 10-minute break, use Stethee® to auscultate and identify the same set of 10 manikin-simulated heart sounds but played in a different sequence to Test 1.
  Interventions: Device: Stethee®; Device: 3MTM Littmann® Classic IIITM

INTERVENTIONS:
Device: Stethee® — Stethee® is a new wireless digital stethoscope.
Device: 3MTM Littmann® Classic IIITM — 3MTM Littmann® Classic IIITM is the conventional stethoscope.

SUMMARY:
The objective of this study is to compare the relative capability of Stethee® (new wireless digital stethoscope) and 3M™ Littmann® Classic III™ (conventional stethoscope) in the identification of manikin-simulated heart sounds by medical doctors. A randomised, non-blinded, two-period crossover, non-inferiority design will be used to compare the acoustic performance of the two stethoscopes. We aim to determine if Stethee® is as effective as 3M™ Littmann® Classic III™ for auscultation of simulated heart sounds, and whether Stethee® could be recommended for use in clinical practice based on a non-inferior comparison with 3M™ Littmann® Classic III™.

DETAILED DESCRIPTION:
This is a randomised, non-blinded, two-period crossover, non-inferiority study. Stethee®, a new wireless digital stethoscope, is designed to minimise ambient noise associated with electronic stethoscopes. To date, its acoustic capability in comparison to the conventional stethoscope in the auscultation of heart sounds is not known. Therefore, it is important that Stethee®'s capability as a stethoscope with sound amplification be evaluated alongside the conventional stethoscope prior to its use in the clinical setting. As acoustic performance is the primary endpoint, a non-inferiority design is proposed to enable the comparison of the mutual functionalities of the two stethoscopes. The rationale for a non-inferiority design is that: (a) electronic stethoscopes have shown a marginal benefit over conventional stethoscopes in terms of acoustic performance; (b) electronic stethoscopes have several functional advantages over conventional stethoscopes: the ability to analyse heart sounds and record heart sounds, the availability of a database for storage of heart sounds for remote analysis; and (c) electronic stethoscopes were rated better than conventional stethoscopes in terms of the overall quality of auscultation.

The relative capability of Stethee® is compared to that of 3M™ Littmann® Classic III™ by the identification of heart sounds simulated by a manikin, which functions as a surrogate patient. A random sample of non-specialist doctors stratified by health centres in Perak, Malaysia, who meet eligibility criteria and provide written consent to participate, will be randomised to initial testing with Stethee® or 3M™ Littmann® Classic III™ to perform cardiac auscultation on a manikin and identify a set of 10 heart sounds. After a 10-minute break, they will repeat the auscultation of the same 10 simulated heart sounds but played in a different sequence with the alternate stethoscope. Following the completion of both tests, the doctors will be asked to complete a questionnaire that asks about their preference for either Stethee® or 3M™ Littmann® Classic III™ with respect to ease of use, audio clarity, and diagnostic accuracy. At the end of the study, answer sheets and preference questionnaires will be collected for grading and analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Non-specialist medical doctors with up to 6 years of working experience post-house officer training
2. Non-specialist medical doctors currently working in the Medical, Paediatric, Anaesthesiology, and Emergency departments of specialist hospitals

Exclusion Criteria:

1. Non-specialist medical doctors who have worked in the Cardiology department for more than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Correctly identified manikin-simulated heart sounds | Measured immediately after the test
  The proportion of correctly identified heart sounds between groups will be compared. The test consist of 10 cardiac conditions (represented by 10 manikin-simulated heart sounds). Subjects (medical doctors) are required to auscultate each heart sound and write the complete answer on the answer sheet. The 'all-or-nothing' marking scheme is used, i.e. answers must exactly match the marking scheme.

SECONDARY OUTCOMES:
User preference for the two stethoscopes | Measured immediately after the test
  User preference for the two stethoscopes with respect to ease of use, audio clarity, and diagnostic accuracy, will be compared between groups. This will be estimated as a proportion preferring Stethee® for each domain.
Difference in the performance between subgroup of doctors from different clinical settings | Measured immediately after the test
  The performance of subgroup of doctors in specialist hospitals and doctors in non-specialist hospitals or primary care clinics will be compared. This will be estimated as a proportion difference of correctly identified heart sounds for each doctor subgroup.
Comparison of the performance of the two stethoscopes in identifying heart sounds of different levels of difficulty | Measured immediately after the test
  The performance of the two stethoscopes in identifying heart sounds of different levels of difficulty (normal, easy, moderately difficult, difficult) will be compared. This is estimated as a proportion difference of correctly identified heart sounds for each type of heart sound.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wei Yin Lim, Pharmacy, Principal Investigator — Clinical Research Centre, Malaysia; Amar Singh HSS, Paediatrics, Principal Investigator — Clinical Research Centre, Malaysia
Locations (1):
- Raja Permaisuri Bainun Hospital, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No